CLINICAL TRIAL: NCT01989429
Title: A Randomized, Double-blind, Parallel Group Phase III Multi-center Trial to Compare Twice Daily Topical Application of M518101, Daivonex® and Vehicle in Patients With Plaque Psoriasis III
Brief Title: Efficacy Study Comparing Topical M518101 and Vitamin D3 in Adult Psoriasis Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Maruho Europe Limited (Industry)
Collaborators: Maruho Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M518101-EU04; 2013-001632-21 (EudraCT Number)
Record Dates: First submitted 2013-10-28; First posted 2013-11-21 (Estimated); Last update posted 2015-12-31 (Estimated); Status verified 2015-12

CONDITIONS: Plaque Psoriasis
Keywords: psoriasis; Vitamin D3; topical; ointments
MeSH Terms: conditions — Psoriasis | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Daivonex (Active Comparator): topical application
  Interventions: Drug: M518101
- vehicle (Placebo Comparator): topical application
  Interventions: Drug: M518101
- M518101 (Experimental): topical application
  Interventions: Drug: M518101

INTERVENTIONS:
Drug: M518101 — 8-week comparative treatment period ( twice daily application) followed by a maximum 8-week period to evaluate time to relapse
  Other Names: vitamin D3; psoriasis treatment

SUMMARY:
M5181 - a novel vitamin D3 analogue - is currently under development for the treatment of plaque psoriasis and is being developed as a topical ointment formulation (M518101)

Clinical and non-clinical studies indicate that M5181 is an effective treatment for plaque psoriasis.

Based on the results of previous phase II trials the phase III trial has been designed to evaluate efficacy and safety of an 8-week treatment period with 50 μg/g M518101 in a larger population of patients with stable plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 18 years or older on the day of signing the informed consent form (ICF)
* Psoriasis patients with up to 20% affected body surface area ( BSA) (not including face or scalp)
* Investigator Global Assessment(IGA) of moderate to severe and who are suitable for topical therapy

Exclusion Criteria:

* Pregnant or lactating females;
* Patients with known allergic reactions, irritations or sensitivity to vitamin D3 derivatives drug hypersensitivity to other components of the investigational products;
* Patients who have been treated with topical steroids, topical immunosuppressive/ immunomodulative drugs, topical vitamin D3 derivative, topical retinoids, anthralin, coal tar (except when used as shampoo) salicylic acid within 14 days of randomization
* Patients, who in the opinion of the investigator, have clinically relevant history or presence of any disease, any other skin disorder, any chronic medical condition which is not well controlled or surgical history which may interfere with the conduct of the trial
* Patients whose calcium test at screening exceed the upper limit of reference range (including serum calcium, albumin, phosphate, parathyroid hormone);
* Patients who have used any study drug (including experimental biologics) and/or participated in any clinical trial within the last 60 days before the day of randomization
* Patients who have been treated with any biologics for their psoriasis within 30 days or 5 half-lives (whichever is longer) of the biologic before the day of randomization the longest documented half-life of the biologic should be used to calculate the 5 half-lives;
* Patients who have been treated with phototherapy (laser, oral steroids, oral retinoid, oral immunosuppressive/immunomodulative drugs, cytostatics, cyclosporine or methotrexate within 30 days of randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 788 (Actual)
Dates: Start 2013-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Severity of psoriasis | 8 weeks
  % reduction in mPASI(modified psoriasis area and severity index) will be measured

SECONDARY OUTCOMES:
Duration of response following 8 week treatment | 8 weeks
  if mPASI is reduced by 50% or more at V7 , patients will be followed up for a further 8 weeks to evaluate time to relapse

CONTACTS AND LOCATIONS:
Overall Officials: D Thaci, Prof.Dr, Principal Investigator — University of Lubeck, Dermatology Department
Locations (6):
- Universitätsklinik für Dermatologie und Venerologie,, Graz, Austria
- DCC "Chaika" EOOD, Varna, Bulgaria
- Universitatsklinikum Schleswig-Holstein, Lübeck, Germany
- Semmelweis Hospital, Miskolc, Csabai Kapu 9-11,, Hungary
- PI Hospital of Lithuanian University of Health Sciences, Kaunas, Lithuania
- CSK MON Wojskowego Instytutu Medycznego, Warsaw, Poland